CLINICAL TRIAL: NCT05427227
Title: A Clinical Study Initiated by Investigator:Prospectively Predict the Efficacy and Explore the Mechanism of Precise Treatment of Gastrointestinal Tumors Based on Peripheral Blood Multi- Omics Liquid Biopsy
Brief Title: Prospectively Predict the Efficacy and Explore the Mechanism of Treatment of Gastrointestinal Tumors Based on Peripheral Multi-omics Liquid Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: CGOG-EV-1002
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Advanced or Late Stage Gastrointestinal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gastrointestinal cancer (GI) patients receiving immunotherapy
  Interventions: Device: EV-array detection
- GI patients receiving anti-HER2 therapy
  Interventions: Device: EV-array detection
- GI patients receiving anti-CLDN18.2 therapy
  Interventions: Device: EV-array detection

INTERVENTIONS:
Device: EV-array detection — Collect peripheral blood sample of 500 GI patients at treatment baseline, every time point response till disease progression.Blood samples will be transferred to central lab to detect certain exosome proteins expression by EV-array.Tumor response evaluation will be performed after two cycles of therapy by CT/MRI based on RECIST.Clinical data, including tumor stage,metastatic organ ,regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
Dynamic multiomics detection of plasma derived exosomes to explore the efficacy and mechanism of anti-HER2, immunotherapy and anti-CLDN18.2 of gastrointestinal cancer.

DETAILED DESCRIPTION:
The investigators will recruit 500 advancer/late-stage gastrointestinal cancer patients.Blood and tumor tissue will be collected at treatment baseline, every time point response till disease progression. All samples will be processed by exosomes proteome detection to explore the efficacy and mechanism of anti-HER2, immunotherapy and anti-CLDN18.2 of gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

* • Having signed informed consent

  * Age:18-80 years old
  * Histologically confirmed GI cancer
  * Unresectable recurrent or metastatic GI cancer
  * Previous neo-adjuvant or adjuvant treatment for GI cancer, if applicable, more than 6 months
  * Measurable disease according to the RECIST criteria
  * Karnofsky performance status ≥70
  * Life expectancy of ≥3 month
  * No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
  * ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
  * Serum albumin level ≥3.0g/dL
  * Serum AKP < 2.5 times ULN
  * Serum creatinine <ULN, and CCr < 60ml/min
  * Bilirubin level < 1.5 ULN
  * WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Previous systemic therapy for metastatic GI cancer

  * Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
  * Allergic constitution or allergic history to protium biologic product or any investigating agents.
  * Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
  * Pregnancy or lactation period
  * Other previous malignancy within 5 year, except non-melanoma skin cancer
  * Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study were enrolled by the Department of gastrointestinal oncology, Peking University Cancer Hospital & Institute for conventional therapy or clinical trials
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Tumor associated proteins expression level of exosomes | Treatment baseline; Up to 2 months from the initial treatment; From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  90 tumor associated proteins' expression level of plasma derived exosomes at treatment baseline, second time point response and disease progression time point will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided